CLINICAL TRIAL: NCT06590090
Title: Phase II, Double-Blind, Placebo-Controlled, Randomized Trial Examining Natrunix in Combination With Methotrexate for the Treatment of Rheumatoid Arthritis
Brief Title: Natrunix in Combination With Methotrexate for Rheumatoid Arthritis Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT067
Record Dates: First submitted 2024-08-22; First posted 2024-09-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 400mg Natrunix + MTX weekly (Experimental): Subjects will receive 400mg Natrunix and MTX weekly
  Interventions: Biological: Natrunix 400 mg; Drug: Methotrexate (MTX)
- Placebo+ MTX weekly (Experimental): Subjects will receive placebo and MTX weekly
  Interventions: Drug: Placebo; Drug: Methotrexate (MTX)

INTERVENTIONS:
Biological: Natrunix 400 mg — The active ingredient of Natrunix is an IgG4 monoclonal antibody indistinguishable from that naturally occurring in an IL-1a-immune healthy human.
  Natrunix is formulated as 200 mg/mL sterile liquid in a stabilizing isotonic formulation buffered to pH 7.0. The product is filled into a 2 mL glass pre-filled syringe suitable for subcutaneous injection. The drug product is formulated and buffered to a neutral body pH of 7.0.
  Other Names: methotrexate
  Arms: 400mg Natrunix + MTX weekly
Drug: Placebo — Placebo is a sterile liquid solution filled into a 2 mL glass pre-filled syringe, suitable for subcutaneous injection, containing the exact same buffer matrix used for Natrunix drug product
  Arms: Placebo+ MTX weekly
Drug: Methotrexate (MTX) — Methotrexate may be administered in pill form by mouth, as liquid by mouth, or by subcutaneous injection.Subjects enrolled in this study should be receiving a stable minimum weekly dose of 10mg. Weekly methotrexate should not exceed 25 mg/week.

SUMMARY:
Approximately 108 subjects will be randomized in 2 arms in 2:1 ratio to receive weekly subcutaneous injections of either 400mg Natrunix + MTX weekly or placebo + MTX weekly for 14 weeks. At the week 14 visit subjects in both arms will undergo a safety follow up visit OR begin receiving biweekly subcutaneous injections of 400mg Natrunix for 14 weeks as part of an Open Label Extension (OLE).

The study will last for a maximum of 33 weeks, including: a screening period of up to 4 weeks, a 14-week double-blinded treatment phase followed by a 14-week open label extension phase and one-week follow-up.

DETAILED DESCRIPTION:
Number of Planned Subjects: Approximately 108 subjects within 2 arms randomized 2:1 [400 mg Natrunix + MTX weekly (n=72) or placebo + MTX weekly arms (n=36)].

Study Duration: The study will last for a maximum of 33 weeks, including: a screening period of up to 4 weeks, a 14-week double-blinded treatment phase followed by a 14-week open label extension phase and one-week follow-up.

Study Design: Subjects will be randomized into the study in a 2:1 ratio to receive weekly subcutaneous injections of either 400mg Natrunix + MTX weekly or placebo + MTX weekly for 14 weeks. At the week 14 visit subjects in both arms will undergo a safety follow up visit OR begin receiving biweekly subcutaneous injections of 400mg Natrunix for 14 weeks as part of an Open Label Extension (OLE).

Subjects will undergo a preliminary assessment for study eligibility. Subjects who meet pre-screening requirements may then provide informed consent to acknowledge understanding of and accept enrollment into the clinical study. Subjects enrolled in the study will be taking concomitant methotrexate, have a diagnosis of moderate to severe RA according to 2010 ACR/EULAR classification criteria and have ≥6 swollen joints (based on DAS28), ≥6 tender joints (based on DAS28) and DAS-ESR > 3.2.

ELIGIBILITY:
Inclusion Criteria:

1. Weight > 40 kg
2. Diagnosis of moderate to severe RA according to 2010 ACR/EULAR classification criteria.
3. Patients must be methotrexate-inadequate responders.

   a. Persistent moderate to severe RA disease activity (i.e., criteria #2 above) despite ongoing treatment with MTX.
4. Meets the following minimum disease activity criteria at screening: ≥6 swollen joints (based on DAS28) and ≥6 tender joints (based on DAS28) and DAS-ESR (Erythrocyte Sedimentation Rate) > 3.2.
5. Subject must be receiving MTX treatment at a dosage of 10-25 mg/week for a minimum of 12 weeks; and be receiving a stable dose of MTX for >4 weeks preceding randomization. Subjects must also be in principle agreement to remain at the pre-randomization stable dose of MTX for the entire duration of the study. Subjects must also be willing to take a minimum of 5 mg folic acid/folinic acid per week for the duration of the study.
6. Subjects must have discontinued all csDMARDs (excluding MTX) for at least 4 weeks or 5 half-lives prior to enrollment, whichever is longer.
7. Subjects taking regular NSAIDs, Acetaminophen, oral corticosteroids (<10mg/day prednisone equivalent), and inhaled corticosteroids must be on a stable dose for 2 weeks prior to enrollment.
8. Subjects must have discontinued high potency opioids (oxycodone, fentanyl, etc.) for at least 4 weeks prior to enrollment.
9. Male or female, at least 18 years of age, willing to provide informed consent, able to attend all clinic visits, comply with study-related procedures and able to understand and complete study-related questionnaires.
10. Patients must provide at least 7 consecutive days of NRS-pain data in the subject's diary prior to the baseline visit. The NRS pain diary should ideally be completed for the 7 days immediately prior to Visit 1 (when the first dose of test drug is administered). Subjects may record more than 7 days of pain records in the diary for their baseline. At least seven consecutive days of pain diary are necessary to be eligible for enrollment in the study.
11. Peripheral blood CD19+ cell count recovery to >10 cells/uL or >1% of total lymphocyte count (Required only for subjects who have received a Rituximab (or anti-CD20 biosimilar) infusion within 12 months prior to enrollment).
12. Female patients of childbearing potential must consent to undergo a serum pregnancy test at enrollment, and urine pregnancy tests at each visit after screening. Women of non-childbearing potential include those considered to have a medical history that indicates that pregnancy is not a reasonable risk, including post-menopausal women and those with a history of hysterectomy or surgically sterilized.
13. In case of female patients of childbearing potential, willingness to use one method of contraception of high efficacy during the entire study period. These methods can include but not limited to hormonal contraceptives, intrauterine devices, condoms, diaphragms, etc.
14. Males participating in this clinical research study should not get a sexual partner pregnant during their participation in this research study as the effect of the study drug on sperm is not known. Male contraception methods can include but are not limited to mechanical methods (e.g., abstinence, non-vaginal intercourse), contemporary methods comprising barrier methods (e.g., spermicide, condom, sponge, diaphragm and cervical cap) and vasectomy.

Exclusion Criteria:

1. History of treatment with Natrunix for any reason.
2. Any active, chronic, or recurrent infections. (e.g., ongoing bacterial, viral, or fungal infection).
3. Comorbid severe psychiatric illness and/or complicated social situations that would limit compliance with study requirements.
4. Patients with a positive result of TB test (QuantiFERON-TB Gold (QFT) at screening unless the patients can present a documentation of completion of TB treatment course by the local Health Department and a clear chest x-ray at enrollment.
5. Patients who have failed more than 1 conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) regimen (excluding Methotrexate monotherapy) due to inefficacy at any point prior to enrollment.
6. Patients who have received any biological therapy including anakinra, rilonacept, canakinumab, adalimumab, certolizumab, etanercept, golimumab, infliximab, abatacept, tocilizumab, sarilumab, and biosimilars at any point prior to enrollment.
7. Treatment with JAK inhibitors at any point prior to enrollment.
8. Patients who have received treatment with Injectable corticosteroids within 8 weeks prior to enrollment.
9. Investigational therapy administered within a time interval less than at least 5 half-lives of the investigational agent prior to the first scheduled day of dosing in this study.
10. Pregnant or breastfeeding patients.
11. Patients with current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within a year prior to enrollment.
12. Uncontrolled heart disease, including NYHA Class III or IV congestive heart failure, ventricular arrhythmia, uncontrolled blood pressure (defined as ≥ 160/100 mm Hg), or unstable angina.
13. Clinically significant laboratory abnormalities, including:

    1. Hemoglobin <9.0 g/dL
    2. White blood cell counts < 4000/mm3
    3. Absolute neutrophil count (ANC) <1500/mm3
    4. Platelet count <100,000/mm3
    5. Absolute lymphocyte count (ALC) <500/mm3
    6. eGFR <45 mL/min
    7. Alanine Aminotransferase (ALT) >1.5x lab upper limit of normal (ULN)
    8. Aspartate Aminotransferase (AST) >1.5x lab upper limit of normal (ULN)
    9. Bilirubin >1.5x lab upper limit of normal (ULN)
14. Major surgery (including joint surgery) within 3 months of baseline.
15. Patients who have suffered severe trauma or fracture within 4 weeks of baseline.
16. Evidence of active hepatitis B, hepatitis C, or HIV infection.

    1. Patients positive for HBsAg and/or positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded.
    2. Patients who are positive for Hepatitis C antibody and negative when the Hepatitis C RNA-PCR assay is performed on a subsequent sample will be eligible to participate. Patients who are positive for Hepatitis C antibody and have a positive result for the HCV when the Hepatitis C RNA-PCR assay is performed on the subsequent sample will not be eligible to participate.
17. Any other concomitant disease, disorder, or condition that could interfere with the interpretation of study endpoints, or the patient's ability to participate in and complete the study, including but not limited to:

    1. Coexisting diseases which are contraindicated for MTX treatment.
    2. Cardiovascular, renal, pulmonary, gastrointestinal, or nervous system disorders that, in the opinion of the principal investigator and/or study medical monitor, make the patient not suitable for enrollment.
    3. Concurrent autoimmune disease excluding Sjogren's syndrome secondary to rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-07-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
ACR 20 response | at 14 weeks from baseline
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.

SECONDARY OUTCOMES:
ACR 50 response rate | at 14 weeks from baseline
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.
Mean change in number of swollen and tender joints based on 66/68-joint count | at 14 weeks from baseline
  Subject's tender and swollen joint will be counted by investigators
Mean change in NRS-pain score | at 14 weeks from baseline
  Subjects will rate the pain score everyday between 7-10pm, where 0 is no pain and 10 is maximum pain
ACR 70 response rate | at 2, 4, 8, 12 and 14 weeks from baseline
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.
ACR 20 response rate | at 2, 4, 8 and 12 weeks from baseline
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.
ACR 50 response rate | at 2, 4, 8 and 12 weeks from baseline
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.
Mean change in HAQ-DI score | at 2, 4, 8, 12 and 14 weeks from baseline
  HEALTH ASSESSMENT QUESTIONNAIRE (HAQ) DISABILITY INDEX (DI): This questionnaire is used in this study which has 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities subjects will be assessed on. In each section, 0 represents without any difficulty and 3 represents task cannot be done at all. In each section, if one question is scored 1 and another 2, then the score for the section is 2. If an aid or device is used or if help is required from another individual, then the minimum score for that section is 2. If the section score is already 2 or more then no modification is made. If any task is not applicable, it can be left blank by the subject.
Mean change in NRS-pain score | at 2, 4, 8 and 12 weeks from baseline
  Subjects will rate the pain score everyday between 7-10pm, where 0 is no pain and 10 is maximum pain
Mean change in RAPID-3 score | at 2, 4, 8, 12 and 14 weeks from baseline
  The RAPID3 (Routine Assessment of Patient Index Data 3) is an index of data set measures to assess disease severity. Each measure is scored 0 to 10, for a total of 30. Higher RAPID3 scores correlate with higher disease severity (>12 = high; 6.1-12 = moderate; 3.1-6 = low; < 3 = remission).
Mean change in the PGA score | at 2, 4, 8, 12 and 14 weeks from baseline
  A patient global assessment (PGA) score is a single question with a 0 to 10 response. Higher scores represent a higher level of disease activity or a worse global health.
Mean change in the EGA score | at 2, 4, 8, 12 and 14 weeks from baseline
  The evaluator global assessment (EGA) score is a single question used to assess how well a patient is doing regarding the status of a disease. This is scored 0-10, higher scores represent worse activity.
Mean change in number of swollen and tender joints based on 66/68-joint count | at 2, 4, 8, and 12 weeks from baseline
  Subject's tender and swollen joint will be counted by investigators
Mean change in the CDAI score | at 2, 4, 8, 12 and 14 weeks from baseline
  The Clinical Disease Activity Index (CDAI) is a composite index for assessing disease activity, it is based on the count of swollen/tender joint count of 28 joints along with patient and evaluator global assessments. The CDAI has a range of 0 -76 and can be classified as: remission (≤2.8), low disease activity (2.9-10), moderate disease activity (10.1-22), and high disease activity (>22).
Mean change in DAS28-ESR score | at 2, 4, 8, 12 and 14 weeks from baseline
  The Disease Activity Score (DAS28) with (Erythrocyte Sedimentation Rate) is a calculator for rheumatoid arthritis that measures disease activity on a scale of 0-10. A higher score indicates more active disease:
  <2.6: Remission 2.6-3.2: Low disease activity 3.2-5.1: Moderate disease activity >5.1: High disease activity
Percentage of patients with Low Disease Activity (DAS-ESR <3.2; CDAI > 2.8 & ≤ 10) | at 2, 4, 8, 12 and 14 weeks from baseline
  The Disease Activity Score (DAS28) with (Erythrocyte Sedimentation Rate) is a calculator for rheumatoid arthritis that measures disease activity on a scale of 0-10. A higher score indicates more active disease.
  The Clinical Disease Activity Index (CDAI) for Rheumatoid Arthritis determines severity of rheumatoid arthritis
Occurence of AEs and SAEs in subjects during the trial | until 28 weeks from baseline
  Subjects will be monitored for any adverse events or serious adverse reactions due to study drug
Any abnormality in Physical examination will be monitored | until 28 weeks from baseline
  Physical examination is the process of evaluating objective anatomic findings through the use of observation, palpation, percussion, and auscultation.
Any clinically significant changes in vital signs from normality will be assessed | until 28 weeks from baseline
  Vital signs are measurements of the body's most basic functions, such as breathing rate, heart rate, body temperature, and blood pressure.
Any abnormal laboratory tests will be monitored | until 28 weeks from baseline
  Laboratory test is a medical procedure that involves testing a sample of blood, urine, or other substance from the body.
ACR 20 response rate | at 22 and 28 OLE weeks
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.
ACR 50 response rate | at 22 and 28 OLE weeks
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.
ACR 70 response rate | at 22 and 28 OLE weeks
  The American College of Rheumatology (ACR) response criteria for rheumatoid arthritis (RA) are used to measure how effective study drug is in this study.
Mean change in number of swollen and tender joints based on 66/68-joint count | at 22 and 28 OLE weeks
  Subject's tender and swollen joint will be counted by investigators
Mean change in NRS-pain score | at 22 and 28 OLE weeks
  Subjects will rate the pain score everyday between 7-10pm, where 0 is no pain and 10 is maximum pain
Mean change in HAQ-DI score | at 22 and 28 OLE weeks
  HEALTH ASSESSMENT QUESTIONNAIRE (HAQ) DISABILITY INDEX (DI): This questionnaire is used in this study which has 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities subjects will be assessed on. In each section, 0 represents without any difficulty and 3 represents task cannot be done at all. In each section, if one question is scored 1 and another 2, then the score for the section is 2. If an aid or device is used or if help is required from another individual, then the minimum score for that section is 2. If the section score is already 2 or more then no modification is made. If any task is not applicable, it can be left blank by the subject.
Mean change in RAPID-3 score | at 22 and 28 OLE weeks
  The RAPID3 (Routine Assessment of Patient Index Data 3) is an index of data set measures to assess disease severity. Each measure is scored 0 to 10, for a total of 30. Higher RAPID3 scores correlate with higher disease severity (>12 = high; 6.1-12 = moderate; 3.1-6 = low; < 3 = remission).
Mean change in the PGA score | at 22 and 28 OLE weeks
  A patient global assessment (PGA) score is a single question with a 0 to 10 response. Higher scores represent a higher level of disease activity or a worse global health.
Mean change in the EGA score | at 22 and 28 OLE weeks
  The evaluator global assessment (EGA) score is a single question used to assess how well a patient is doing regarding the status of a disease. This is scored 0-10, higher scores represent worse activity.
Mean change in the CDAI score | at 22 and 28 OLE weeks
  The Clinical Disease Activity Index (CDAI) is a composite index for assessing disease activity, it is based on the count of swollen/tender joint count of 28 joints along with patient and evaluator global assessments. The CDAI has a range of 0 -76 and can be classified as: remission (≤2.8), low disease activity (2.9-10), moderate disease activity (10.1-22), and high disease activity (>22).
Mean change in DAS28-ESR score | at 22 and 28 OLE weeks
  The Disease Activity Score (DAS28) with (Erythrocyte Sedimentation Rate) is a calculator for rheumatoid arthritis that measures disease activity on a scale of 0-10. A higher score indicates more active disease:
  <2.6: Remission 2.6-3.2: Low disease activity 3.2-5.1: Moderate disease activity >5.1: High disease activity
Percentage of patients with Low Disease Activity (DAS-ESR <3.2; CDAI > 2.8 & ≤ 10) | at 22 and 28 OLE weeks
  The Disease Activity Score (DAS28) with (Erythrocyte Sedimentation Rate) is a calculator for rheumatoid arthritis that measures disease activity on a scale of 0-10. A higher score indicates more active disease.
  The Clinical Disease Activity Index (CDAI) for Rheumatoid Arthritis determines severity of rheumatoid arthritis
Assessment of Maximum Plasma Concentration | at baseline (pre-treatment) until week 14
  Blood samples will be collected from subjects. Maximum Plasma Concentration (Cmax) measurement of Natrunix will be performed in all enrolled participants.
Number of participants with Anti-Drug Antibodies | at baseline (pre-treatment) until week 14
  Blood samples will also be used to test for the presence of treatment emergent anti-drug antibodies (ADA) against Natrunix. XBiotech has developed an ELISA method to perform quantitative and qualitative measurements of ADA.
ECG QTc interval | until 28 weeks from baseline
  An electrocardiogram (ECG or EKG) is a non-invasive test that records the cardiac electrical activity. QTc(ms) value will be collected along with a clinical interpretation. A normal QTc interval on an ECG, is generally considered to be between 350 and 450 milliseconds (ms) for men and 360 to 460 ms for women. Any abnormalities in ECG will be recorded during study from baseline.

IPD SHARING:
Plan to Share IPD: Undecided